CLINICAL TRIAL: NCT04367831
Title: Intermediate or Prophylactic-Dose Anticoagulation for Venous or Arterial Thromboembolism in Severe COVID-19: A Cluster Based Randomized Selection Trial (IMPROVE-COVID)
Brief Title: Intermediate or Prophylactic-Dose Anticoagulation for Venous or Arterial Thromboembolism in Severe COVID-19
Acronym: IMPROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sahil A. Parikh, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS8980
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Venous Thromboses; Arterial Thrombosis
Keywords: COVID-19; coronavirus; anticoagulation
MeSH Terms: conditions — COVID-19; Venous Thrombosis; Coronavirus Infections | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention arm: intermediate-dose anticoagulation (Experimental): If estimated glomerular filtration rate (eGFR) ≥ 30 mL/min: enoxaparin 1mg/kg subcutaneous (SC) daily or unfractionated heparin infusion at 10 units/kg/hour with goal anti-Xa 0.1-0.3 U/mL.
  If eGFR <30 mL/min or acute kidney injury or CRRT: Unfractionated heparin infusion at 10 units/kg/hour (minimum 500 units/hour if CRRT) with goal anti-Xa 0.1-0.3 U/mL
  Interventions: Drug: Heparin Infusion; Drug: Enoxaparin/Lovenox Intermediate Dose
- Control arm: prophylaxis (Active Comparator): Prophylactic dose anticoagulation (per Columbia University Irving Medical Center (CUIMC) Guidelines):
  If eGFR ≥30 mL/min (stable kidney function):
  1. BMI < 40 kg/m2: Enoxaparin 40 mg SC daily
  2. BMI 40 - 50 kg/m2: Enoxaparin 40 mg SC q12h
  3. BMI > 50 kg/m2: Enoxaparin 60 mg SC q12h
  If eGFR < 30 mL/min or acute kidney injury:
  1. 50-120 kg: Unfractionated heparin 5000 units SC q8h
  2. >120 kg: Unfractionated heparin 7500 units SC q8h
  If CRRT: Unfractionated heparin infusion pre-filter at 500 units/hour
  Interventions: Drug: Enoxaparin Prophylactic Dose; Drug: Heparin SC

INTERVENTIONS:
Drug: Enoxaparin Prophylactic Dose — Prophylactic dose anticoagulation (per Columbia University Irving Medical Center (CUIMC) Guidelines):
  If eGFR ≥30 mL/min (stable kidney function):
  1. BMI < 40 kg/m2: Enoxaparin 40 mg SC daily
  2. BMI 40 - 50 kg/m2: Enoxaparin 40 mg SC q12h
  3. BMI > 50 kg/m2: Enoxaparin 60 mg SC q12h
  Other Names: Lovenox
  Arms: Control arm: prophylaxis
Drug: Heparin Infusion — Unfractionated heparin infusion at 10 units/kg/hour with goal anti-Xa 0.1 -0.3U/mL.
  Other Names: Heparin
  Arms: Intervention arm: intermediate-dose anticoagulation
Drug: Heparin SC — Unfractionated heparin at 5000-7500 units subcutaneous (SC) every 8 hours.
  Other Names: Heparin
  Arms: Control arm: prophylaxis
Drug: Enoxaparin/Lovenox Intermediate Dose — If estimated glomerular filtration rate (eGFR) ≥ 30 mL/min: enoxaparin 1mg/kg subcutaneous (SC) daily.
  Other Names: Lovenox
  Arms: Intervention arm: intermediate-dose anticoagulation

SUMMARY:
This study is being conducted to assess the effectiveness of intermediate versus prophylactic doses of anticoagulation (blood thinners) in patients critically ill with COVID-19 in the intensive care units (ICUs) throughout the hospital. Anticoagulation is part of the patient's usual standard of care but determining the dose of anticoagulation is based on physician preference. The investigators are conducting this study (a randomized trial with adaptive design employing cluster randomization) with the support of all of the ICUs to collect data in order to determine what should be the standard of care in terms of anticoagulation in these critically ill patients. The patients care will not be altered other than the choice of anticoagulation (both approved and used throughout the hospital as standard of care) based on the ICU bed they are assigned. Patient data will be collected until discharge.

DETAILED DESCRIPTION:
Hemostatic, biomarker, and inflammatory changes are common in severe manifestations of coronavirus disease 2019 (COVID-19).Such factors, as well as the bedridden status and critical illness may constitute a prothrombotic milieu, predisposing to venous and arterial thrombosis. However, the optimal antithrombotic regimen for patients with COVID-19, especially those with severe disease, remains uncertain and is currently an area of active clinical interest. Prophylactic-dose anticoagulation is generally recommended for acutely ill hospitalized patients. However, given the hemostatic abnormalities of severe COVID-19 illness, it is unknown whether more intensive anticoagulation is preferred to reduce the risk of thrombotic events, potentially mitigating microvascular and macrovascular thrombi and even disseminated intravascular coagulation (DIC). Further, the risks of therapeutic dose anticoagulation must be weighed against the bleeding risks inherent to this approach. To address this critical gap in knowledge in an area of clinical equipoise, the investigators plan to conduct a cluster-randomized trial in patients admitted to intensive care units (ICUs) in a large volume academic medical center to select the best anticoagulation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 by reverse transcription polymerase chain reaction (RT-PCR)
* New admission to eligible CUIMC ICUs within 5 days

  * Transfer from nonparticipating to participating ICU is eligible if otherwise meets eligibility criteria.
  * Patients transferred between participating ICUs will maintain initial treatment assignment.
  * Patients not on therapeutic anticoagulation and who were already admitted to participating ICU within 5 days of trial initiation are additionally eligible.

Exclusion Criteria:

* Weight under 50kg
* Contraindication to anticoagulation in the opinion of the treating clinician including

  * overt bleeding
  * platelet count <50,000
  * Bleeding Academic Research Consortium (BARC) major bleeding in the past 30 days
  * Gastrointestinal (GI) bleeding within 3 months
  * history of intracranial hemorrhage
  * Ischemic stroke within the past 2 weeks
  * craniotomy/major neurosurgery within the past 30 days
  * cardiothoracic surgery within the past 30 days
  * intra-abdominal surgery within 30 days prior to enrollment
  * Head or spinal trauma in the last months
  * History of uncorrected cerebral aneurysm or arteriovenous malformation (AVM)
  * Intracranial malignancy
  * Presence of an epidural or spinal catheter
  * Recent major surgery within the last 14 days
  * Decrease in hemoglobin >3 g/dL over the last 24 hours
  * Allergic reaction to anticoagulants (e.g. Heparin Induced Thrombocytopenia) as documented in the electronic health records. Extracorporeal membrane oxygenation (ECMO) support or other mechanical circulatory support.
* Severe chronic liver dysfunction (history of portosystemic hypertension (HTN), esophageal varices, or Child-Pugh class C or above or similar Model For End-Stage Liver Disease (MELD) scores), abnormality in liver function tests (aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin) 5 times greater than upper normal limit.
* A history of congenital bleeding diatheses or anatomical anomaly that predisposes to hemorrhage (e.g. hemophilia, hereditary hemorrhagic telangiectasia)
* Treating physician preference for therapeutic anticoagulation
* Enrollment in other concurrent trials related to anticoagulant or antiplatelet therapy
* Existing treatment with therapeutic anticoagulation during the previous 7 days of hospitalization prior to ICU admission (e.g. for venous thromboembolism (VTE), atrial fibrillation, mechanical valve, etc).
* Do-not-resuscitate (DNR) /do-not-intubate (DNI) or comfort measures only (CMO) orders prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, Study Chair — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- [Derived] Levi M, Thachil J, Iba T, Levy JH. Coagulation abnormalities and thrombosis in patients with COVID-19. Lancet Haematol. 2020 Jun;7(6):e438-e440. doi: 10.1016/S2352-3026(20)30145-9. Epub 2020 May 11. No abstract available. PMID 32407672

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Intensive Care Units
Groups:
- Intervention Arm: Intermediate-dose Anticoagulation: If estimated glomerular filtration rate (eGFR) ≥ 30 mL/min: enoxaparin 1mg/kg subcutaneous (SC) daily or unfractionated heparin infusion at 10 units/kg/hour with goal anti-Xa 0.1-0.3 U/mL.
  If eGFR <30 mL/min or acute kidney injury or CRRT: Unfractionated heparin infusion at 10 units/kg/hour (minimum 500 units/hour if CRRT) with goal anti-Xa 0.1-0.3 U/mL
  Heparin Infusion: Unfractionated heparin infusion at 10 units/kg/hour with goal anti-Xa 0.1 -0.3U/mL.
  Enoxaparin/Lovenox Intermediate Dose: If estimated glomerular filtration rate (eGFR) ≥ 30 mL/min: enoxaparin 1mg/kg subcutaneous (SC) daily.
- Control Arm: Prophylaxis: Prophylactic dose anticoagulation (per Columbia University Irving Medical Center (CUIMC) Guidelines):
  If eGFR ≥30 mL/min (stable kidney function):
  1. BMI < 40 kg/m2: Enoxaparin 40 mg SC daily
  2. BMI 40 - 50 kg/m2: Enoxaparin 40 mg SC q12h
  3. BMI > 50 kg/m2: Enoxaparin 60 mg SC q12h
  If eGFR < 30 mL/min or acute kidney injury:
  1. 50-120 kg: Unfractionated heparin 5000 units SC q8h
  2. >120 kg: Unfractionated heparin 7500 units SC q8h
  If CRRT: Unfractionated heparin infusion pre-filter at 500 units/hour
  Enoxaparin Prophylactic Dose: Prophylactic dose anticoagulation (per Columbia University Irving Medical Center (CUIMC) Guidelines):
  If eGFR ≥30 mL/min (stable kidney function):
  1. BMI < 40 kg/m2: Enoxaparin 40 mg SC daily
  2. BMI 40 - 50 kg/m2: Enoxaparin 40 mg SC q12h
  3. BMI > 50 kg/m2: Enoxaparin 60 mg SC q12h
  Heparin SC: Unfractionated heparin at 5000-7500 units subcutaneous (SC) every 8 hours.
Period: Overall Study
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Started | 46; 4 Intensive Care Units | 48; 4 Intensive Care Units
Completed | 46; 4 Intensive Care Units | 48; 4 Intensive Care Units
Not Completed | 0; 0 Intensive Care Units | 0; 0 Intensive Care Units

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (12.2) | 63.2 (11.5) | 62.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 36 | 67
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 33 | 66
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Patients Who Were Alive and Without Venous/Thrombotic Events in ICU
Description: Composite of being alive and without clinically-relevant venous or arterial thrombotic events at discharge from ICU (without transfer to another ICU or palliative care unit/hospice) or at 30 days (if ICU duration lasted 30 days or longer).
Time Frame: Discharge from ICU or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
Participants | 28 | 31

2. Secondary Outcome: Total Number of Patients With Clinically Relevant Venous or Arterial Thrombotic Events in ICU
Description: Composite of being alive and with clinically relevant venous or arterial thrombotic events at discharge from ICU (without transfer to another ICU or palliative care unit/hospice) or at 30 days (if ICU duration lasted 30 days or longer).
Time Frame: Discharge from hospital or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
Participants | 15 | 18

3. Secondary Outcome: ICU Length of Stay
Description: Length of stay measured in days.
Time Frame: Discharge from ICU, up to 36 days
Measure: Mean (Full Range); unit: days
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
days | 23 [1 to 36] | 26 [1 to 34]

4. Secondary Outcome: Total Number of Patients With the Need for Renal Replacement Therapy in the ICU
Description: The impact of intermediate-dose anti-coagulation compared with prophylactic anti-coagulation on rates of acute kidney injury and renal recovery in the ICU will be measured with the total number of patients who need of renal replacement therapy in the ICU.
Time Frame: Discharge from ICU or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
Participants | 11 | 15

5. Secondary Outcome: Total Number of Patients With Major Bleeding in the ICU
Description: Major bleeding will be assessed by BARC criteria (> BARC 3), also explored by International Society on Thrombosis and Haemostasis (ISTH) and Thrombolysis in Myocardial Infarction (TIMI) criteria.
Time Frame: Discharge from ICU or 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
Participants | 5 | 5

6. Secondary Outcome: Hospital Length of Stay
Description: Length of stay measured in days.
Time Frame: Discharge from ICU, up to 36 days
Measure: Mean (Full Range); unit: days
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
Number analyzed (Participants) | 46 | 48
days | 17.78 [1 to 36] | 17.73 [1 to 34]

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Intervention Arm: Intermediate-dose Anticoagulation | Control Arm: Prophylaxis
All-Cause Mortality (participants affected / at risk) | 10/46 | 11/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 15/46 | 12/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm: Intermediate-dose Anticoagulation (N=46) | Control Arm: Prophylaxis (N=48)
Venous Thromboembolism (Vascular disorders) | 5 | 6
Actionable Line Thrombosis (Vascular disorders) | 6 | 7
CVVH Filter Thrombosis (Vascular disorders) | 3 | 1
Acute Kidney Injury (Renal and urinary disorders) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04367831/Prot_SAP_000.pdf